CLINICAL TRIAL: NCT01738893
Title: Bioequivalence Study Between Two Medications for Administration of Oral Gabapentin in 300 mg Capsules in Healthy Volunteers
Brief Title: Bioequivalence Study of 300 mg Gabapentin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 116850
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Epilepsy
Keywords: Gabapentin; Bioequivalence; Pharmacokinetics; Mexico
MeSH Terms: conditions — Epilepsy | interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (test)/ B (reference) (Experimental): initial administration of test and cross-over to reference
  Interventions: Drug: Gabapentin 300 mg
- B (reference/ A (test) (Experimental): initial administration of reference and cross-over to test
  Interventions: Drug: Gabapentin 300 mg

INTERVENTIONS:
Drug: Gabapentin 300 mg — Test product
  Other Names: Darbetin®; Laboratorios Dermatologicos Darier
Drug: Gabapentin 300 mg — Reference product
  Other Names: Nerotin®; Pfizer

SUMMARY:
The objective of this study was to confirm if two formulations of gabapentin (capsules) are bioequivalent.

Test product was Darbetin® 300 mg (Laboratorios Dermatológicos Darier) and reference product Nerotin® 300 mg (Pfizer). One capsule was the single dosage.

The study was prospective, open-label, randomized, crossover, single dose, with 02 treatments, 02 sequences and 02 periods, under fasting conditions.

The population was composed of 26 healthy volunteers, both genders, adults between 18-55 years.

The comparative bioavailability of the two formulations was evaluated based in statistical comparisons of relevant pharmacokinetic parameters, obtained from data of drug concentrations in blood.

ELIGIBILITY:
Inclusion Criteria:

Males 18-55 years. Healthy based on comprehensive medical history, lab tests, Chest x-ray, Electrocardiogram, negative tests for Hepatitis B and C, and HIV. Negative urine doping test. BMI 19-26.5 kg/m2. Lab test in normal range +/- 10%. Blood pressure 139-90/89-50, heart rate 100-55, respiratory rate 24-17, temperature 37.5-35 °C. Non-smoking at least for 10 hrs before study. Written informed consent. Women must be not pregnant, nor breast-feeding.

-

Exclusion Criteria:

Hypersensitivity to study medication or other related drug. History of cardiovascular, renal, hepatic, metabolic, gastrointestinal, neurologic, endocrine, hematopoietic, psychiatric or organic condition.

Requiring any drug interfering with minocycline pharmacokinetics. Exposed to inducers or inhibitors of hepatic enzymes. Intake of possible toxic drugs 30 days before study. Intake of any drug 14 days or 7 half-lives before study. Hospitalization or severe disease 60 days before study. Receiving investigational drug out of study center 30 days before study. Blood loss or blood donation =>450 ml 60 days before study. Recent history of drug abuse including alcohol. Intake of xanthine containing products 10 hrs before study. Intake of grapefruit juice or hot-spice 10 hrs before study.

-

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2011-01-14 (Actual); Primary Completion 2011-01-22 (Actual); Study Completion 2011-01-22 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (CMAX) of drug gabapentin | 0.0, 0.50, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 8.0, 10.0, 12.0, and 24.0 postdosage
  Pharmacokinetics
Area under the plasma concentration versus time curve (AUC) of gabapentin | 0.0, 0.50, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 8.0, 10.0, 12.0, and 24.0 postdosage
  Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- See also: Results for study 116850 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116850?search=study&search_terms=116850#rs